CLINICAL TRIAL: NCT00011960
Title: A Randomized Phase II Comparison Of Two Cisplatin-Paclitaxel Containing Chemoradiation Regimens In Resected Gastric Cancers
Brief Title: Chemotherapy and Radiation Therapy With or Without Fluorouracil in Treating Patients With Cancer of the Stomach Who Have Undergone Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-G-0114; CDR0000068464
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Paclitaxel; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cisplatin and paclitaxel use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Cisplatin and paclitaxel may make the tumor cells more sensitive to radiation therapy and may kill any tumor cells remaining after surgery.

PURPOSE: Randomized phase II trial to study the effectiveness of cisplatin, paclitaxel, and radiation therapy with or without fluorouracil in treating patients who have stage IB, stage IIB, or stage IIIB stomach cancer that has been removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 2-year disease-free survival in patients with resected stage IB-IIIB gastric cancer treated with cisplatin, paclitaxel, and radiotherapy with or without fluorouracil vs therapy in the adjuvant arm of the intergroup adjuvant protocol 0116 (RTOG 90-18). (Arm I closed to accrual as of 6/18/03.)
* Compare the safety and success of these regimens vs therapy in the intergroup adjuvant study.
* Compare the toxic effects of these regimens vs therapy in the adjuvant arm of the intergroup study.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor stage (T1-2 vs T3 vs T4) and by number of involved lymph nodes (none vs 1-3 vs 4 or more). Patients are randomized to one of two treatment arms. (Arm I closed to accrual as of 6/18/03.)

* Arm I (closed to accrual as of 6/18/03): Patients receive fluorouracil IV continuously and cisplatin IV over 1 hour on days 1-5 and 29-33 and paclitaxel IV continuously on days 1 and 29.

At 3-4 weeks after completion of chemotherapy, patients receive radiotherapy once daily and fluorouracil IV continuously on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive paclitaxel IV over 3 hours on days 1, 8, 15, 22, and 29.

* Arm II: Patients receive paclitaxel IV over 3 hours and cisplatin IV over 1 hour on days 1 and 29.

At 3-4 weeks after completion of chemotherapy, patients receive radiotherapy once daily and paclitaxel IV continuously on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive cisplatin IV over 1 hour on days 1, 8, 15, 22, and 29.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 94 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IB-IIIB adenocarcinoma of the stomach or gastroesophageal junction having undergone potentially curative resection of primary tumor

  * No more than 8 weeks since primary tumor resection
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC (white blood cell count) at least 4,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine amino transferase) no greater than 2.5 times upper limit of normal

Renal:

* BUN(blood urea nitrogen)less than 30 mg/dL
* Creatinine no greater than 1.4 mg/dL
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No active angina or myocardial infarction within the past 6 months
* No history of significant ventricular arrhythmia requiring medication with antiarrhythmics
* No history of clinically significant conduction system abnormality

Other:

* No concurrent serious infection that is uncontrolled or would preclude study participation
* No nonmalignant medical illness that is uncontrolled or would preclude study participation
* No psychiatric disorders that would preclude study participation
* No other active malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No clinically significant hearing loss
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the treatment field

Surgery:

* See Disease Characteristics

Other:

* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paul Kelsen, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (69):
- United States (69):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Baptist Hospital of Miami, Miami, Florida
  - Alexian Brothers Cancer Care Center, Elk Grove Village, Illinois
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Wayne Memorial Hospital, Inc., Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital - Summa Health System, Akron, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - St. Charles Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital - ProMedica Health System, Sylvania, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - University of Washington Medical Center, Seattle, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Schwartz GK, Winter K, Minsky BD, Crane C, Thomson PJ, Anne P, Gross H, Willett C, Kelsen D. Randomized phase II trial evaluating two paclitaxel and cisplatin-containing chemoradiation regimens as adjuvant therapy in resected gastric cancer (RTOG-0114). J Clin Oncol. 2009 Apr 20;27(12):1956-62. doi: 10.1200/JCO.2008.20.3745. Epub 2009 Mar 9. PMID 19273696
- [Result] Schwartz GK, Winter K, Minsky B, et al.: A randomized phase II trial comparing two paclitaxel (P)-cisplatin (C) containing chemoradiation (CRT) regimens as adjuvant therapy in resected gastric cancer (RTOG 0114). [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1069, S169, 2006.